CLINICAL TRIAL: NCT02219321
Title: Lidocaine Infusion for Chronic Pain in Opioid Dependent Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Enas Kandil, Asistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 062014-002
Record Dates: First submitted 2014-08-14; First posted 2014-08-18 (Estimated); Results first posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Chronic Pain
Keywords: Pain, Opioid dependence, Lidocaine infusion
MeSH Terms: conditions — Chronic Pain; Pain; Opioid-Related Disorders | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine infusion (Active Comparator): A continuous intravenous infusion of lidocaine
  Interventions: Drug: Lidocaine infusion
- Saline infusion (Placebo Comparator): A continuous intravenous infusion of saline
  Interventions: Drug: Saline infusion

INTERVENTIONS:
Drug: Lidocaine infusion — Lidocaine intravenous 2mg/kg initial bolus over 5 minutes followed by a continuous intravenous infusion of lidocaine at a rate of 2mg /kg /hour for 4 hours
  Other Names: Intravenous lidocaine
  Arms: Lidocaine infusion
Drug: Saline infusion — A continuous intravenous infusion of saline at the same volume with lidocaine infusion for 4 hours
  Other Names: Isotonic Sodium Chloride
  Arms: Saline infusion

SUMMARY:
Prescription drug abuse represents a major healthcare problem, with treatment costs reaching billions of dollars annually in the United States alone. Today opioids are commonly prescribed for chronic non-cancer pain and are only partially effective for short-term pain relief. Whereas opioids are initially part of the solution for pain, it eventually often turns to be a problem in patient with chronic pain. Long-term treatment with opioids can be complicated by development of tolerance, dependency, addiction, abnormal pain sensitivity, hormonal changes, and immune modulation. Unfortunately, the chronic use of anti-inflammatory drugs is associated with a marked increase in adverse effects.

The purpose of this study is to determine whether systemic administration of lidocaine provides effective pain relief in opioid dependent chronic pain patients. Investigators intend to demonstrate that lidocaine infusion can improve pain relief and physical function in opioid dependent patients, thus improving compliance and patient satisfaction, which may potentially help wean patients off narcotics. The long-term goal of this proposal is to decrease opioid dependence in chronic pain patients by using lidocaine infusion.

DETAILED DESCRIPTION:
There is a significant disconnect between the escalating healthcare problem of opioid use for chronic pain, and the development of novel therapeutic strategies. A plausible strategy is to interrupt the vicious cycle of pain, inflammation and hyperesthesia is using highly efficacious non-opioid drugs that do not require chronic administration, such as lidocaine. Lidocaine is FDA approved local anesthetic, class 2 antiarrhythmic with analgesic, antihyperalgesic and anti-inflammatory properties without rewarding and addictive properties. Intravenous lidocaine has been utilized since 1943 for a large spectrum of pain conditions. Lidocaine also has been shown to significantly reduce circulating inflammatory cytokines production. Investigators propose that systemic administration of lidocaine will decrease the intensity, duration of pain in opioid dependent chronic pain patients. The long-term goal of this proposal is to decrease opioid dependence in chronic pain patients by using lidocaine infusion. The central hypothesis is that lidocaine infusion decreases the intensity of pain in opioid dependent chronic pain patients.

Primary outcome: To determine the short-term effect of lidocaine infusion on the intensity of pain in opioid dependent chronic pain patients.

Secondary outcome1: Determine the duration of pain relief after lidocaine infusion in opioid dependent chronic pain patients. Investigators hypothesize that lidocaine infusions will have a long lasting Visual Analog Pain (VAS) score improvement that will extend beyond the time of infusion.

This intermediate and long-term pain relief will be demonstrated by measuring both VAS pain scores 3 times a day for 3 weeks and by the reduction in daily opioid use by 25%.

Secondary outcome2: Determine the effect of lidocaine infusion on opioid induced hyperalgesia. Lidocaine infusion may decrease cytokine levels both acutely after infusion as compared to baseline, as well as at the end of 1 week after infusion.

STUDY DESIGN AND POPULATION: Forty opioid dependent patients will be randomized in a double blind parallel placebo control study to investigate the effects of lidocaine on neuropathic pain. Patients who meet the inclusion criteria will receive Initial laboratory work-up prior to infusion date. Each patient will receive a Hepatic panel, CBC, and Chemistry and baseline cytokine levels (IL1b) as well as a baseline Cold Pressor Test (CPT) and then will be randomized to either receive lidocaine or placebo.

Study Intervention: Lidocaine intravenous 2mg/kg initial bolus over 5 minutes followed by a continuous intravenous infusion of lidocaine at a rate of 2mg /kg /hour for 4 hours versus saline of same volume and duration.

Duration of the study: Patient will be followed for 3 weeks after the lidocaine infusion.

Monitoring during infusion: Heart rate, blood pressure, EKG, oxygen saturation, and any potential side effects as sedation, circumoral numbness, metallic taste in the mouth will be continuously monitored and recorded every 15 minutes (standard monitoring and recording time in recovery area) as well as pain scores. After completion of infusion patient will be further monitored for another 2 hrs and then discharged after meeting standard discharge criteria according to Aldrete scoring system.

Discharge instruction: Patients will be asked to decrease their daily opioid dose by 25%. Patients will receive a one-week supply of a short acting opioid as a rescue medication. Patients will be asked to use the rescue medication if pain is moderate to severe for the first day after infusion. If no improvement in pain despite allowable short acting medication as reported on first day post infusion follow up phone call, patient will be asked to resume their usual long acting opioid dose. Each patient will receive a pain diary sheet where they will record their daily visual analogue pain scores 3 times a day as well as their daily opioid dose plus over the counter analgesic requirements as NSAIDS and acetaminophen. Patients will follow up every week till study completion, where pain diary, over the counter and rescue pain medications will be assessed.

Outcome Measures:

1. Visual Analog Pain (VAS) Scores
2. Serum interleukin Ib level
3. CPT
4. Daily opioid use

Subject Safety and Data Monitoring:

All subjects will be carefully assessed prior to participation in the studies, including medical history, laboratory tests, and examination by a board-certified physician (Dr. Kandil). Subjects with medical problems that would increase risk for participation will be excluded from the study.

During the infusion patient's vital signs: heart rate, blood pressure, EKG, oxygen saturation, and any potential side effects as sedation, circumoral numbness, metallic taste in the mouth will be continuously monitored and recorded every 15 minutes as well as pain scores.

All lidocaine/saline infusions will be supervised by Dr. Enas Kandil, an anesthesiologist. Dr. Kandil or a nurse will be in attendance during throughout the infusion. Heart rate, including EKG rhythm strip, will be monitored continuously throughout the infusion and blood pressure will be obtained every 15 minutes and more frequently if indicated. If the participants' hemodynamics (heart rate, blood pressure) change by more than 20% (typically a consequence of cardiac arrhythmias) the infusion will be stopped. The more serious toxic effects of lidocaine (e.g. unconsciousness, confusion, convulsions, respiratory arrest) are preceded by numbness of the tongue, lightheadedness, visual disturbances and muscle twitching; infusions will be terminated if the subject reports of any of these latter signs or symptoms. A checklist of signs and symptoms will be obtained every 15 minutes. Subjects will be observed for at least two hours (approximately one half-life of lidocaine) following the cessation of lidocaine (or saline) infusion. Dr. Kandil must approve discharge for all participants on the infusion study day.

Lidocaine labels carry warnings and precautions for use in patients with various cardiac conditions, notably conduction abnormalities (e.g., heart block, QT prolongation). Cardiac conditions will be identified by EKG, medical history and physical exam. Participants with any medical history of cardiac disease (e.g. myocardial infarction, congestive heart failure, cardiac arrhythmia) or an abnormal EKG (including any arrhythmia, heart block, QT prolongation) will be excluded.

Women with a positive pregnancy test or who report unprotected heterosexual sex since their previous menses will not receive an infusion. Women with a positive pregnancy test will be referred for appropriate care. Subjects will be observed for at least two hours (approximately one half-life of lidocaine) following the cessation of lidocaine (or saline) infusion. All participants will receive a 24-hour call-in number to contact research staff in the advent of problems.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old -Patient currently on stable dose of opioids for more than six months period -
* Patients with Chronic uncontrolled neuropathic pain with documented pain score > or = 4 despite opioids
* Not currently abusing opioids or other illicit drugs as demonstrated by history and negative urine toxicology screen
* Patient agrees to come to all follow up visits at 1, 2, and 3 week following infusion
* Having baseline/screening EKG

Exclusion Criteria:

* Individuals meeting DSM-V dependence criteria for alcohol, benzodiazepine, CNS stimulant, marijuana or other drug of abuse.
* Hepatic dysfunction as determined by history and physical or clinical significant lab.
* Cardiac arrhythmias including heart block and QT prolongation as determined by history or baseline EKG.
* Subject has inability to understand and cooperate with study procedures or provide informed consent.
* Subject has history of intolerance or allergic reaction to lidocaine.
* Subject has history of seizures.
* Raynaud's disease
* Renal impairment as determined by clinically significant labs.
* Women of childbearing age who either have:

  1. A positive pregnancy test
  2. Unprotected heterosexual sex since their previous menses or;
  3. Not currently using and/or willing to use a medically approved form of contraception (e.g., birth control pill).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2015-05-14 (Actual); Study Completion 2019-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enas Kandil, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Parkland Health Hospital System, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lidocaine Infusion | Saline Infusion
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine Infusion | Saline Infusion | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Continuous [Mean (Full Range); unit: years] | 51 [51 to 51] | 57 [50 to 64] | 55 [50 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 0

OUTCOME MEASURES:

1. Primary Outcome: Intensity of Pain
Description: Visual Analog Pain Scores on a scale of 0 to 10 (0=no pain and 10=worst pain)
Time Frame: Immediately after continuous 4-hours Intravenous lidocaine infusion
Population: Chronic pain patients with opioid precription
Measure: Median (Full Range); unit: units on a scale 0 to 10
Arm/Group | Lidocaine Infusion | Saline Infusion
Number analyzed (Participants) | 1 | 2
units on a scale 0 to 10 | 8 [7 to 8] | 3 [0 to 3]

2. Secondary Outcome: Withdrawal Time (Seconds)
Description: The time to withdraw at the Cold Pressor Task immediately after 4-hours intravenous continuous lidocaine infusion
Time Frame: Immediately after Lidocaine Infusion
Measure: Mean (Full Range); unit: seconds
Arm/Group | Lidocaine Infusion | Saline Infusion
Number analyzed (Participants) | 1 | 2
seconds | 61 [61 to 61] | 41.5 [24 to 59]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected during lidocaine infusion and 2 hours immediately after the infusion and during 3-weeks follow-up period
Arm/Group | Lidocaine Infusion | Saline Infusion
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes